CLINICAL TRIAL: NCT04912401
Title: A Prospective Study With Induction Dosing Period Followed by a Maintenance Dosing Period to Evaluate the Efficacy and Safety of Etanercept （Yi Sai Pu) in Chinese Patients With Moderate-to-Severe Psoriasis
Brief Title: the Efficacy and Safety of Etanercept （Yi Sai Pu) in Chinese Patients With Moderate-to-Severe Psoriasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Xiaoyong Man, Principal Investigator, Head of Dermatology, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: 2020-915
Record Dates: First submitted 2021-03-01; First posted 2021-06-03 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Psoriasis; Etanercept
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, open-label, one-arm study. The study aims to assess the efficacy and safety of Etanercept therapy which help guide the clinical practice in real-world settings.

ELIGIBILITY:
Inclusion Criteria:

1.18 to 75 years of age 2.Moderate to severe chronic psoriasis, BSA≥3% 3.Duration of psoriasis≥6 months 4.Patients must be candidate for systemic therapy or phototherapy 5.No contradiction to Etanercept 6.Informed consent must be obtained 7.For female, ß-hCG test is negative and contraception is accepted

Exclusion Criteria:

1. Diagnosis of pustular psoriasis, erythroderma psoriasis or drug-induced psoriasis
2. Having severe infections, including hepatitis, HIV and tuberculosis
3. No live vaccines 12 weeks before enrollment, through the study and 1 year after the last dose of Etanercept
4. Having significant allergies to biological agents
5. Having the previous experience of biologics
6. Having a history of malignancy
7. Having contradictions to Etanercept
8. Refusal of contraception
9. Having serious or unstable/uncontrolled illnesses

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe psoriasis (PASI>3) and bio-naive
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-04 (Actual); Primary Completion 2025-12-04 (Estimated); Study Completion 2025-12-04 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients achieving PASI75 at week 12 | 12 weeks
  PASI75: 75% improvement from baseline in the Psoriasis Area and Severity Index (PASI) scores. PASI includes desquamation, erythema, and plaque induration/infiltration.

SECONDARY OUTCOMES:
Percentage of patients achieved PASI90 at week 12 | 12 weeks
  PASI90: 90% improvement from baseline in the Psoriasis Area and Severity Index (PASI) scores.
Percentage of patients achieved PASI90 at week 24 | 24 weeks
  PASI90: 90% improvement from baseline in the Psoriasis Area and Severity Index (PASI) scores.
Percentage of patients achieved PASI90 at week 36 | 36 weeks
  PASI90: 90% improvement from baseline in the Psoriasis Area and Severity Index (PASI) scores.

CONTACTS AND LOCATIONS:
Locations (40):
- China (40):
  - 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - First Affiliated Hospital, Zhejiang Medical University, Hangzhou
  - Hang Zhou First People's Hospital, Hangzhou
  - Hang Zhou Third People's Hospital, Hangzhou
  - Hospital of dermatology of Xiaoshan, Hangzhou
  - Sir Run Run Shaw Hospital of College of Medicine of Zhejiang University, Hangzhou
  - the People Hospital of Zhejiang Province, Hangzhou
  - Xiaoshan Hospital, Hangzhou
  - Yuhang Fifth People's Hospital, Hangzhou
  - Zhejiang Hospital of Traditional Chinese Medicine, Hangzhou
  - Changxing Dermatology Hospital prevention and Treatment, Huzhou
  - Chinese 72 Hospital, Huzhou
  - Hospital of dermatology of Zhejiang Province, Huzhou
  - Huzhou Central Hospital, Huzhou
  - Huzhou First Hospital, Huzhou
  - the People Hospital of Changxing, Huzhou
  - Jiaxing First Hospital, Jiaxing
  - Rongjun Hospital of Zhejiang Province, Jiaxing
  - Tongxiang Dermatology Hospital prevention and Treatment, Jiaxing
  - Hospital of dermatology of Yiwu, Jinhua
  - Jinhua Central Hospital, Jinhua
  - Jinhua Fifth Hospital, Jinhua
  - the People Hospital of Dongyang, Jinhua
  - Lishui Central Hospital, Lishui
  - the People Hospital of Lishui, Lishui
  - Ningbo Chinese Medical Hospital, Ningbo
  - Ningbo First Hospital, Ningbo
  - Ningbo Sixth Hospital, Ningbo
  - Quzhou Chinese Medical Hospital, Quzhou
  - the People Hospital of Quzhou, Quzhou
  - Shangyu of Chinese Medical Hospital, Shaoxing
  - Shaoxing Central Hospital, Shaoxing
  - Shaoxing Third Hospital, Shaoxing
  - the People Hospital of Shaoxing, Shaoxing
  - Taizhou Central Hospital, Taizhou
  - Wenling Chinese Medical Hospital, Taizhou
  - the First Affiliated Hospital of Wenzhou medical university, Wenzhou
  - the People Hospital of Cangnan, Wenzhou
  - Wenzhou Chinese Medical Hospital, Wenzhou
  - Wenzhou Combinational Hospital of Chinese and Western Medicine, Wenzhou

IPD SHARING:
Plan to Share IPD: No